CLINICAL TRIAL: NCT03671980
Title: Feasibility and Acceptability of an Inflammatory Bowel Disease Self-management Website and Home Faecal Calprotectin Monitoring After Treatment De-escalation
Brief Title: IBD Self-management Website and Home Faecal Calprotectin Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHM MED1269
Record Dates: First submitted 2017-06-13; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Self-care
Keywords: Calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-intervention (Experimental): 30 participants using a self-management website and home faecal calprotectin smartphone monitoring instead of usual outpatient follow up as a means of managing their inflammatory bowel disease for 6 months after stopping an IBD medication.
  Interventions: Other: My Medical record website

INTERVENTIONS:
Other: My Medical record website — Website comprising patient records, blood and other test results, useful information on IBD, and messaging service to communicate with IBD team, plus home smartphone faecal calprotectin monitoring.

SUMMARY:
6 month exploratory feasibility study to assess if a combination of MyMedicalRecord supported self-management website and a home faecal calprotectin smartphone testing kit is a feasible and acceptable means for patients to monitor for signs of relapse after treatment de-escalation.

DETAILED DESCRIPTION:
IBD can be challenging to manage as disease flares are often unpredictable and rarely coincide with scheduled outpatient appointments. Websites are a novel way of assisting patients to take more control over monitoring and managing symptoms and have been shown to improve outcomes in some chronic diseases. The My Medical Record (MyMR) webiste was developed to help patients learn about IBD, access test results, monitor symptoms, and manage their medications, with email support from the IBD team.

The use of home faecal calprotectin monitoring will also be explored. This marker of IBD activity is normally performed in hospital laboratories and becomes elevated before the onset of clinical symptoms of an IBD flare. New technologies enable patients to perform the test at home with the aid of a smartphone application.

A 6 month exploratory feasibility study will be conducted to assess if a combination of MyMR and a home faecal testing kit is a feasible and acceptable means for patients to monitor their illness. Their use will be targeted to patients who have recently stopped (or reduced) a treatment for IBD, as up to 50% of these patients may have a disease flare within a year.

Interventions

* Clinic appointments Study participants will not be required to attend any routine outpatient follow up appointments for the 6 month study period, after which they will be reviewed by a member of the IBD team.
* Questionnaires and interviews Partcipants will receive questionnaires and a sample will also undergo interviews to explore their views regarding the website and stool test.
* Website

Participants will be encouraged to use all functions of the website at least monthly:

1. Secure email messaging service
2. IBD educational material
3. Stool, nutritional and flare journals
4. Blood and test results
5. Faecal calprotectin monitoring - monthly testing (or sooner if symptoms of a flare-up) using QuantonCal home faecal calprotectin smartphone application. Participants will test and monitor their FC levels monthly. The results will be overseen by the IBD team who will make contact within a week in the event of abnormal results if the participant has not already done so.

   * Blood tests All participants will have a routine blood test at 0 and 6 months. Those taking azathioprine, mercaptopurine and methotrexate should continue regular blood monitoring (minimum of 3 monthly FBC, U&E, LFT and CRP) as usual practice. Participants will be provided with blood test results and explanations of their significance via MyMR. The results will be overseen by the IBD team who will make contact within a week in the event of abnormal results if the patient has not already done so.
   * Safety Patients can contact the IBD team the email messaging service at any time for advice and support.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years currently under secondary care outpatient follow up for IBD
* Diagnosed with IBD at least one year prior to study enrolment (to ensure patients are familiar with their disease and treatments)
* Stopped or reduced the dose of one or more treatments for IBD (for any reason) within the last 8 weeks
* Able to understand English and provide written consent.
* Own, or have regular (at least weekly) access to a smartphone +/- personal computer with internet

Exclusion Criteria:

* Inability to read, understand informed consent
* Inability to use a smartphone
* Likely requirement of IBD surgery within the study period
* Ileostomy
* Pregnancy or planned pregnancy within next 6 months
* Terminal illness with limited (< 1year) life expectancy
* Current participation in another IBD research study
* Any reason, in the opinion of the investigators, which is likely to make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Faecal calprotectin testing completion rates | 6 months
  Number of patients completing monthly faecal calprotectin testing
MyMR website usage | 6 months
  Number of patients logging in to MyMR website at least monthly

SECONDARY OUTCOMES:
Recruitment | 6 months
  Number of patients recruited per month
IBD email contact | 6 months
  Number of email messaging contacts per patient to IBD specialist nursing team
IBD flareline calls | 6 months
  Number of IBD flareline telephone calls per patient to IBD specialist nursing team
IT support contact | 6 months
  Number of IT support email contacts per patient
Questionnaire response rates | 6 months
  Response rates to pre-and post-study questionnaires
Retention rate | 6 months
  Study retention rate (target 80%). Study retention will be defined as successful completion of at least 5 out of 7 home faecal calprotectin tests, with no periods without login to website of greater than 3 consecutive months.
Calprotectin levels | 6 months
  Mean faecal calprotectin levels at 0, 4, 8, 12, 16, 20, and 24 weeks.
IBD-Control | 6 months
  Mean IBD-Control scores at 0, 4, 8, 12, 16, 20, and 24 weeks
SIBDQ | 6 months
  Mean quality of life (SIBDQ) scores at 0 and 26 weeks
IBD knowledge | 6 months
  Mean IBD knowledge scores (CC-KNOW) at 0 and 26 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided